CLINICAL TRIAL: NCT03532594
Title: Algorithmic Protamine Dosing for Reversal of Heparin After Cardiopulmonary Bypass (PRODOSE)
Brief Title: Algorithmic Protamine Dosing for Reversal of Heparin After Cardiopulmonary Bypass
Acronym: PRODOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Austin Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P02337
Record Dates: First submitted 2018-04-26; First posted 2018-05-22 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Heart Diseases; Cardiovascular Diseases
Keywords: Protamine; Heparin Antagonists; Cardiopulmonary Bypass
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The randomisation ratio will be 1:1 in the first instance but the trial uses an adaptive design and an interim analysis will be conducted after 100 patients have been randomised.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Other): At the conclusion of cardiopulmonary bypass, protamine administration will be undertaken at surgical request. For patients in the control group, protamine will be dosed on a 1:1 ratio according to the total dose of heparin initially required to establish a therapeutic activated clotting time (ACT) (i.e. if 30,000 IU were required prior to initiating cardiopulmonary bypass, then the protamine dose will be 300mg).
  Interventions: Procedure: Standard Care
- Algorithm (Experimental): For patients in the intervention group, protamine will be administered according to the PRODOSE algorithm, which has been incorporated into an Excel spread sheet for ease of use (Microsoft Corporation).
  Interventions: Procedure: PRODOSE Algorithm

INTERVENTIONS:
Procedure: PRODOSE Algorithm — Protamine administered according to PRODOSE algorithm
  Arms: Algorithm
Procedure: Standard Care — Protamine administered according to Standard Care
  Arms: Standard Care

SUMMARY:
The PRODOSE trial is investigating a bespoke pharmacokinetic algorithm that calculates a tailored dose of protamine, required after cardiopulmonary bypass to reverse the action of heparin, based on individual patients and their actual bypass time.

The PRODOSE trial aims to demonstrate that the algorithm can be used to define a protamine dose that will more reliably return coagulation parameters to pre-heparin levels as well as decreasing the risk of post-operative bleeding and transfusion.

The trial aims to recruit 200 patients who will be randomised to either a bespoke or standard dose of protamine. The randomisation ratio will be 1:1 in the first instance but the trial uses an adaptive design and an interim analysis will be conducted after 100 patients have been randomised. The randomisation ratio could then be updated after the interim analysis to favour a superior arm whilst preserving statistical power levels.

DETAILED DESCRIPTION:
Open-heart surgery is routinely conducted using a heart-lung machine. In order to conduct operations involving heart-lung machines a patient's coagulation system needs to be reliably suppressed to avoid clot formation. Clot in the extracorporeal circuit generally has fatal consequences.

In the vast majority of cases (>99%) the desired suppression of the blood clotting system is achieved by administering heparin. Although relatively short acting, with a half-life of about 150min for a full adult dose, heparin needs to be reversed after weaning from the heart-lung machine in order to avoid catastrophic bleeding post-operatively.

Heparin reversal is achieved by using protamine. This drug is derived from salmon sperm and is generally safe to use. However, in a reasonable number of cases it can have severe side effects, ranging from dangerous hypotension to high blood pressure in the lung circulation with adequately oxygenate the patient. Severe anaphylactic reactions have also been described. There is also increasing evidence that inadequately high doses of protamine may lead to an increased bleeding tendency.

There is controversy about the right dosing of protamine. Traditionally a pragmatic and empirical '1:1' formula is used reversing 100 Units of heparin with 1mg of protamine. This dosing regime does not take the decay of heparin during the time spent on the heart-lung machine into account and potentially exposes patients to unnecessarily high doses of protamine.

The research team was previously able to demonstrate in a pilot project that using a pharmacokinetic algorithm, which takes heparin decay into account, can reduce the protamine dose given to patients without increased bleeding or transfusion requirements.

The team have continued to develop this algorithm into a 2 compartmental model and are seeking to test the hypothesis that using the new formula can reduce patients' risk of the unwanted side-effects of protamine by reducing its dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective cardiac surgery

Exclusion Criteria:

* Emergency surgery
* Age < 18 years
* Known or suspected coagulopathy or platelet dysfunction
* Adenosine diphosphate (ADP)-receptor antagonists within 7 days of surgery (clopidogrel, ticlopidine, prasugrel)
* Total body weight > 130kg
* End stage renal failure requiring dialysis
* Plan for severe hypothermia (< 28°C) or deep hypothermic circulatory arrest
* Complex cardiac surgery (redo sternotomy, surgery on the thoracic aorta [excluding root])
* Transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Return to normal coagulation after cessation of cardiopulmonary bypass and reversal of heparin | 3 minutes post-protamine administration after cessation of cardiopulmonary bypass.
  Kaolin Thrombelastography (TEG) r-time

SECONDARY OUTCOMES:
Blood loss | 4 hours post-surgery
  Intercostal drain output
Blood products usage | 24 hours post-surgery
  Use of blood products

CONTACTS AND LOCATIONS:
Overall Officials: Florian Falter, FRCA, Principal Investigator — Royal Papworth Hospital NHS Foundation Trust; Lachlan Miles, FRCA, Principal Investigator — Austin Health
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miles LF, Burt C, Arrowsmith J, McKie MA, Villar SS, Govender P, Shaylor R, Tan Z, De Silva R, Falter F. Optimal protamine dosing after cardiopulmonary bypass: The PRODOSE adaptive randomised controlled trial. PLoS Med. 2021 Jun 7;18(6):e1003658. doi: 10.1371/journal.pmed.1003658. eCollection 2021 Jun. PMID 34097705